## **Adult Consent Form**

## Study of the Golimumab Exposure-Response Relationship using Serum Trough Levels

## **GO-LEVEL**

Participant Identification Number for this trial:

| _ | | | _ | |
|----------|-----|----|------|-----|
| D | 200 | ar | ch | er: |
| $\Gamma$ | -55 | aı | UI I | CI. |

| | | | Ple | ase initial box |
|---|---|---|---|---|
| 1. | | ort 1/cohort 2 (delete as applicable) informing the study. I have had the opportunity to contain answered satisfactorily. | | |
| 2. | • • • • | is voluntary and that I am free to withdra my medical care or legal rights being af | • | |
| 3. | may be looked at by individuals from | s of my medical notes and data collected<br>om the NHS Trust and Sponsor, where it<br>sion for these individuals to have access | is relevant to my taking | 9 |
| 4. | . I understand that the anonymised data generated as part of this study will be made available to researchers in the scientific community, including scientists from the pharmaceutical companies who have supported this study, after its completion. | | | |
| 5. | . I understand that laboratory results (blood and stool tests) will be made available to my treating team to help with the management of my condition. | | | |
| 6. | I agree to part of my blood sample | being stored anonymously for use in fut | ure research. | |
| 7. | 7. I agree to take part in the above study. | | | |
| lam | e of participant | Date | Signature | |
| am | e of person taking consent | Date | Signature | nd St Thomas' NHS |

Adult Consent Form (IRAS: 194917) GO-LEVEL Oct 2017 Version 2.1

When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes.

Local contact number: 02071882499